CLINICAL TRIAL: NCT02035033
Title: The Relationship Between Calcium and Cardiac Calcium Scoring
Brief Title: The Relationship Between Ca Intake , Blood Level of Ca, PTH, TSH, Vitamin D, and Urine Ca, P and Cardiac Calcium Scoring
Acronym: TSHPTHCA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Nariman Saba Khazan, Head of Endocrinology Department - Lin, Carmel Medical Center
Other Study IDs: CMC-13-0003-CTIL
Record Dates: First submitted 2013-11-09; First posted 2014-01-14 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Disorders of Phosphorus and Calcium Metabolism

STUDY DESIGN:
Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- low calcium supplement: low calcium supplement
- Calcium intake 500-1000 mg per day: Calcium intake 500-1000 mg per day
- Calcium intake above 1000 mg per day: Calcium intake above 1000 mg per day

SUMMARY:
Osteoporosis (op) is a disorder of bone characterized by reduced mineral density and bone mass. The first step in the prevention and treatment of Op is ensuring adequate intake of calcium and vitamin D . While calcium supplementations clearly slow bone loss in both sexes,their effects on fracture risk are less certain. In contrast to the above a recent randomized, placebo controlled trial in 1471 postmenopausal women (mean age 74) reported in the BMJ (2 February 2008) found an increased rate of vascular events in healthy older women receiving calcium supplementation. The mechanism is not clear .we are trying to identify a possible correlation between calcium intake and calcium cardiac scoring .

DETAILED DESCRIPTION:
BACKGROUND:

1. Osteoporosis (op) is a disorder of bone characterized by reduced mineral density and bone mass. The first step in the prevention and treatment of Op is ensuring adequate intake of calcium and vitamin D . While calcium supplementations clearly slow bone loss in both sexes,(1,2) their effects on fracture risk are less certain.(3,4)
2. Experimental data suggest that . vitamin D 25 affects cardiac muscle directly; controls PTH secretion, regulates the rennin-angiotensin - aldosterone system, and modulates the immune system.(5) Vitamin D deficiency has been associated with hypertension; several types of vascular disease and heart failure.
3. Evidence suggests that high calcium intake might protect against vascular disease.

There is evidence that calcium intake might impact on serum lipid concentrations.(6) There is also evidence that calcium supplementation reduces blood pressure,(7) and that CV mortality is lower in hard water areas.(8)

In contrast to the above a recent randomized, placebo controlled trial in 1471 postmenopausal women (mean age 74) reported in the BMJ (2 February 2008) found an increased rate of vascular events in healthy older women receiving calcium supplementation.

Outcome measures were assesed over 5 years and included death, myocardial infarction, , stroke, transient ischaemic attack and development of angina pectoris.A composite end point of major adverse events (MACE= major advrse cardiac events) included myocardial infarction, stroke, or sudden death. MACE was also more common in the calcium group (101 events in 69 women v 54 events in 42 women, P=0.008). Adjudicated myocardial infarction was more common in the calcium group (24 events in 21 women v 10 events in 10 women, relative risk 2.12, 95% confidence interval 1.01 to 4.47).For stroke the relative risk was 1.37 (0.83 to 2.28) and the rate ratio was 1.45 (0.88 to 2.49). The authors concluded that calcium supplementation in healthy postmenopausal women is associated with upward trends in cardiovascular event rates and that this potentially detrimental effect should be balanced against the likely benefits of calcium on bone. (9) Possible mechanisms: The finding of an adverse trend in vascular events with calcium supplementation is not necessarily surprising, since calcium supplements acutely elevate serum calcium levels possibly accelerating vascular calcification, which is predictive of vascular event rates. Multiple observational studies have shown that cardiac event rate increases markedly over several years of follow-up with increasing levels of CAC(Coronary artery calcium) independently of conventional risk factors. CAC scoring has been advocated asa screening test for coronary disease risk in individuals at intermediate risk for coronary events

AIMS of current study: To define the relationship between calcium in the diet and supplementation to the level of TSH : PTH; vitamin D; creatinine in blood; calcium and Phosphor in blood and urine and the calcium score in the coronary blood vessels .

Methods:

Prospective study One center study includes Carmel hospital ;Line clinic and Zvolon clinic. Collaboration between the radiologic department in Carmel hospital and the endocrine department in Line and Zolon.

Includes 500 participants how recent or planned cardiac CT in the Carmel hospital.

The subject will sign an informed consent before the collection of blood tests for calcium, phosphor, creatinin, vitamin D, and PTH , TSH, urine tests for calcium if they don't have a recent tests(three month) in the OPHEQ .

Questionnaire. -

Inclusion criteria:

Recent or planned coronary artery calcium scoring performed at Carmel Hospital With or without simultaneously performed cardiac CT angiography.

Male and Female. Aged 50-80 years. Hebrew speakers

Exclusion criteria:

Below age 50 years. Above age 80 years. Previous cardiac surgery . Inadequate cardiac CT study

End point:

Correlation between calcium score and the level of VIT D,PTH;TSH in the blood Calcium phosphor in blood and urine and calcium in diet and supplementation.

Statistical analysis:

Standard statistical analysis techniques SPSS 14 (T TEST, ANOVA, Spearman&Pearson correlation, will used in order to find the correlation between calcium score and blood levels of the above.

Bibliography :

1. Randomized controlled trial of calcium supplementation in healthy, non osteoporotic, older men.

   Reid IR; Ames R; Mason B; Reid HE; Bacon CJ; Bolland MJ; Gamble GD; Grey A; Horne A Arch Intern Med. 2008 Nov 10;168(20):2276-82.
2. Randomized controlled trial of calcium in healthy older women. Reid IR; Mason B; Horne A; Ames R; Reid HE; Bava U; Bolland MJ; Gamble GD Am J Med. 2006 Sep;119(9):777-85.
3. Use of calcium or calcium in combination with vitamin D supplementation to prevent fractures and bone loss in people aged 50 years and older: a meta-analysis.

   Tang BM; Eslick GD; Nowson C; Smith C; Bensoussan A Lancet. 2007 Aug 25;370(9588):657-66.
4. Reid ,I.R.,Bolland ,M.J& Gery ,A Effect of calcium supplementation on hip fractures. Osteoporosis International 19 ,1119-1123.
5. Rammos G,Tseke P,Ziakka S. vitamin D,the rennin-angiotensin system,and insulin resistance . Int Urol Nephrology.2008 ;40:419-26.
6. Reid IR, Mason B, Horne A, Ames R, Clearwater J, Bava U, et al. Effects of calcium supplementation on serum lipid concentrations in normal older women: a randomized controlled trial. Am J Med 2002;112:343-
7. Griffith LE, Guyatt GH, Cook RJ, Bucher HC, Cook DJ. The influence of dietary and nondietary calcium supplementation on blood pressure-an updated metaanalysis of randomized controlled trials. Am J Hypertens 1999;12:84
8. Dawson EB, Frey MJ, Moore TD, McGanity WJ. Relationship of metal metabolism to vascular disease mortality rates in Texas. Am J Clin Nutr 1978;31:1188-97
9. Mark J Bolland, research fellow1, P Alan Barber, senior lecturer1, Robert N Doughty, associate professor1, Barbara Mason, research officer1, Anne Horne, research fellow1, Ruth Ames, research officer1, Gregory D Gamble, research fellow1, Andrew Grey, associate professor1, Ian R Reid, professor1 Vascular events in healthy older women receiving calcium supplementation: randomized controlled trial BMJ 2008;336:262-266 (2 February), doi:10.1136/bmj.39440.525752.BE (published 15 January 2008 ontrolled trial.

ELIGIBILITY:
Inclusion Criteria:

Male and Female. Aged 50-80 years. Hebrew speakers -

Exclusion Criteria:

- Below age 50 years. Above age 80 years. Previous cardiac surgery . Inadequate cardiac CT study

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: participants how recent or planned cardiac CT in the Carmel hospital.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-12 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
The safety of calcium intake for heart | 2 years frame

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Peled, Prof., Study Chair — Clalit Health Services